CLINICAL TRIAL: NCT00692913
Title: A Phase III (Phase V Program), Open-Label, Randomized, Referred-Care-Controlled, Clinical Trial to Evaluate the Efficacy and Safety of MK -0217A/Alendronate Sodium-70 mg/Vitamin D3 5600 I.U. Combination Tablet on Vitamin D Inadequacy in the Treatment of Osteoporosis in Postmenopausal Women
Brief Title: A Study to Test the Effect of MK0217A on Vitamin D Inadequacy in Postmenopausal Women With Osteoporosis (0217A-262)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0217A-262; 2007_653
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Cholecalciferol

ARMS (2):
- FOSAVANCE 5600 (Experimental): alendronate sodium (+) cholecalciferol
  Interventions: Drug: FOSAVANCE 5600 (Alendronate Sodium (+) cholecalciferol); Dietary Supplement: Calcium Supplement 500 mg
- Referred-Care Model (Other): Usual treatment for osteoporosis chosen and prescribed by patients' own physicians.
  Interventions: Other: Referred-Care Model

INTERVENTIONS:
Drug: FOSAVANCE 5600 (Alendronate Sodium (+) cholecalciferol) — FOSAVANCE 5600 international units (IU)(Alendronate Sodium 70 mg/Vitamin D 5600 IU) combination tablet once weekly for 6 months (Week 26) during the base period and an additional 6-month extension period (Week 52).
  Arms: FOSAVANCE 5600
Dietary Supplement: Calcium Supplement 500 mg — Calcium supplied locally by the investigator (containing 500 mg
  calcium supplement) daily for 52 weeks (unless the patient's dietary intake of
  calcium exceeds 1000 mg per day).
  Arms: FOSAVANCE 5600
Other: Referred-Care Model — Usual treatment for osteoporosis chosen and prescribed by patients' own physicians for 6 months (Week 26) during the base period and an additional 6-month extension period (Week 52).
  Arms: Referred-Care Model

SUMMARY:
A study designed to see if the study drug will increase blood levels of vitamin D, bone mineral density (BMD), improve biochemical markers of bone turnover, and reduce the number of falls as compared to women receiving standard care for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 65 years or older
* Diagnosed with osteoporosis (Bone Mineral Density (BMD) T-score <= -2.5 at spine or hip) or prior fragility fracture BMD T-score <=-1.5 in at least one of the anatomic sites including lumbar spine, total hip, and femoral neck sites
* Postmenopausal
* Low levels of vitamin D as measured 25-hydroxyvitamin D
* Has fallen at least once within the past 12 months

Exclusion Criteria:

* Unable to stand or sit upright for at least 30 minutes
* Has a bone disorder other than osteoporosis
* Contraindication to the use of FOSAVANCE

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 515 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ralston SH, Binkley N, Boonen S, Kiel DP, Reginster JY, Roux C, Chen L, Rosenberg E, Santora A; FOCUS-D (FOSAVANCE vs. Standard Care-Use and Study of Vitamin D) Trial. Randomized trial of alendronate plus vitamin D3 versus standard care in osteoporotic postmenopausal women with vitamin D insufficiency. Calcif Tissue Int. 2011 Jun;88(6):485-94. doi: 10.1007/s00223-011-9482-4. Epub 2011 Apr 11. PMID 21479913

RESULTS

PARTICIPANT FLOW:
Groups:
- FOSAVANCE 5600: Alendronate Sodium 70 mg/Vitamin D 5600 I.U. combination tablet once weekly plus a daily 500 mg elemental calcium supplement.
- Referred-Care: Usual treatment for osteoporosis chosen and prescribed by patients' own physicians.
Period: Overall Study
Arm/Group | FOSAVANCE 5600 | Referred-Care
Started | 257 | 258
Completed | 228 | 228
Not Completed | 29 | 30
Not completed — Adverse Event | 8 | 4
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSAVANCE 5600 | Referred-Care | Total
Number analyzed (Participants) | 257 | 258 | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (5.3) | 72.9 (5.9) | 72.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257 | 258 | 515
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Levels of 25-hydroxyvitamin D Below 20 ng/mL at Week 26
Description: Percentage of participants with serum levels of 25-hydroxyvitamin D below
  20 nanograms/milliliter (ng/mL) after 26 weeks of treatment with FOSAVANCE 5600 once weekly versus Referred-Care in postmenopausal women with osteoporosis and at increased risk of falls.
Time Frame: Week 26
Population: Full Analysis Set Population (FAS) included participants who took at least one dose of study therapy during the entire treatment period of FOSAVANCE 5600 or who were
  assigned to receive regular care and had data reported at least once post-randomization during the entire study period, and had efficacy measurements during the entire study period.
Measure: Number; unit: Percentage of Participants
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 221 | 216
Percentage of Participants | 8.6 | 31.0
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p < 0.001, Regression, Logistic; The logistic regression model was adjusted by baseline 25-hydroxyvitamin D (25(OH)D) level stratum, age, and region; Odds Ratio (OR) = 0.20, 95% CI [0.12 to 0.35]

2. Secondary Outcome: Percent Change From Baseline at Week 26 in N-Telopeptides of Type 1 Collagen to Urine Creatinine Ratio
Description: N-Telopeptides of Type 1 Collagen to Urine Creatinine Ratio (NTx) is a urine biochemical marker of bone resorption and measured in nanomoles (nmol) Bone Collagen Equivalents (BCE)/millimoles (mmol) creatinine. The percent change was calculated as: [100 * ((Week 26/Baseline)-1)]. The greater the percent decrease from baseline, the greater the response to therapy.
Time Frame: Baseline and Week 26
Population: Per-Protocol Population: excluded participants due to important deviations from the protocol that may substantially affect the results of the primary efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 216 | 226
Percent Change | -57.06 [-60.19 to -53.68] | -47.36 [-51.23 to -43.18]
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; The model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Difference in Least-squares means = -9.70, 95% CI [-14.49 to -4.93]

3. Secondary Outcome: Percent Change From Baseline at Week 26 in Bone-Specific Alkaline Phosphatase
Description: Bone-Specific Alkaline Phosphatase (BSAP) is a serum biochemical marker of bone formation and measured in micrograms/Liter (mcg/L). The percent change was calculated as: [100 * ((Week 26/Baseline)-1)]. The greater the percent decrease from baseline, the greater the response to therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 223 | 237
Percent Change | -46.67 [-49.32 to -43.88] | -39.60 [-42.60 to -36.44]
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; The model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Difference in Least-squares mean = -7.07, 95% CI [-10.95 to -3.20]

4. Secondary Outcome: Percentage of Participants With Serum Levels of 25-hydroxyvitamin D Below 20 ng/mL at Week 52
Description: Percentage of participants with serum levels of 25-hydroxyvitamin D below
  20 ng/mL after 52 weeks of treatment (6 month extension study) with FOSAVANCE 5600 once weekly versus Referred-Care in postmenopausal women with osteoporosis and at increased risk of falls.
Time Frame: Week 52
Population: The FAS population included participants who took at least one dose of study therapy during the entire treatment period of FOSAVANCE 5600 or who were assigned to receive regular care and had data reported at least once post-randomization during the entire study period, and had efficacy measurements during the entire study period.
Measure: Number; unit: Percentage of Participants
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 212 | 203
Percentage of Participants | 11.3 | 36.9
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p < 0.001, Regression, Logistic; The logistic regression model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Odds Ratio (OR) = 0.21, 95% CI [0.13 to 0.35]

5. Secondary Outcome: Percent Change From Baseline in Lumbar Spine and Total Hip Bone Mineral Density
Description: Bone Mineral Density (BMD) as measured by Dual Energy X-Ray Absorptiometry (DEXA) and measured in g/cm^2 was obtained at baseline (visit 1) and Week 52 (visit 13) or at early study discontinuation visit. The percent change was calculated as: [100 * ((Week 52/Baseline)-1)]. The greater the percent change from baseline, the greater the response to therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 227 | 219
Percent Change
  Lumbar Spine (n= 226/ n=219) | 4.92 [4.17 to 5.66] | 3.91 [3.16 to 4.66]
  Total Hip (n=227/ n=218) | 2.22 [1.65 to 2.79] | 1.40 [0.83 to 1.97]
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p = 0.047, Traditional Longitudinal data analysis; The model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Least Squares Mean Difference = 1.01, 95% CI [0.01 to 2.00] — FOSAVANCE minus Referred-Care. Analysis was for Lumbar Spine
Statistical Analysis 2: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p = 0.035, Traditional Longitudinal data analysis; The model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Least Squares Mean Difference = 0.82, 95% CI [0.06 to 1.58] — FOSAVANCE minus Referred-Care. Analysis was for Total Hip

6. Secondary Outcome: Falls Per Participant
Description: Number of falls per participant was measured.
  The fall event rate during the study period was defined as the number of adjudicated falls during the study period divided by the total patient-years in the study. Each participant was to be in the study for approximately one year.
  In order to guide and standardize all procedures during the fall adjudication process, a Standard Operating Procedure for Fall Adjudication was created by the
  SPONSOR and served as a guideline to standardize operational procedures for fall adjudication.
Time Frame: Up to Week 52
Population: Intent-to-Treat (ITT) population included all randomized participants within the treatment group to which they were randomized regardless of whether or not a participant may have dropped out in the base or continued into the extension study.
Measure: Mean (Standard Deviation); unit: Number of Falls
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 257 | 258
Number of Falls | 0.51 (1.53) | 0.45 (0.80)
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p = 0.675, Zero-Inflated Poisson Regression; Adjusted by the terms for treatment, baseline 25(OH) D level stratum, age, and region and offset variable of log (total patient-years in the study); Difference of falls (falls/patient-year) = 0.03, 95% CI [-0.12 to 0.19], Standard Error of Mean 0.08

7. Secondary Outcome: Percent Change From Baseline at Week 52 in N-Telopeptides of Type 1 Collagen to Urine Creatinine Ratio
Description: NTx is a urine biochemical marker of bone resorption and measured in nanomoles (nmol) Bone Collagen Equivalents (BCE)/millimoles (mmol) creatinine. The percent change was calculated as: [100 * ((Week 52/Baseline)-1)]. The greater the percent decrease from baseline, the greater the response to therapy.
Time Frame: Baseline and Week 52
Population: Per-Protocol Population: excluded patients due to important deviations from the protocol that may substantially affect the results of the primary efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 216 | 227
Percent Change | -58.42 [-61.58 to -54.99] | -50.07 [-54.01 to -45.79]
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p = 0.001, Longitudinal Data Analysis Model; The model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Difference in Least Squares Means = -8.35, 95% CI [-13.19 to -3.54]

8. Secondary Outcome: Percent Change From Baseline at Week 52 in Bone-Specific Alkaline Phosphatase
Description: BSAP is a serum biochemical marker of bone formation and measured in micrograms/Liter (mcg/L). The percent change was calculated as: [100 * ((Week 52/Baseline)-1)]. The greater the percent decrease from baseline, the greater the response to therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | FOSAVANCE 5600 | Referred-Care
Number analyzed (Participants) | 223 | 237
Percent Change | -51.21 [-53.79 to -48.48] | -43.13 [-46.18 to -39.91]
Statistical Analysis 1: Comparison: FOSAVANCE 5600 vs Referred-Care; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; The model was adjusted by baseline 25-hydroxyvitamin D level stratum, age, and region; Difference in Least Squares Mean = -8.07, 95% CI [-11.94 to -4.21]

ADVERSE EVENTS:
Description: FOSAVANCE 5600 group: participants who took at least 1 dose were included (254 out of 257 patients). All patients randomized in the referred-care group were included regardless of whether they took 1 dose of therapy as prescribed by their physicians.
Arm/Group | FOSAVANCE 5600 | Referred-Care
Serious Adverse Events (participants affected / at risk) | 25/254 | 29/258
Other Adverse Events (participants affected / at risk) | 61/254 | 70/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSAVANCE 5600 (N=254) | Referred-Care (N=258)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 1 (2)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
Electromechanical Dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Eye Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacterial Diarrhoea (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subacute Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Facial Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Unresponsive to Stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Vascular Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis Superficial (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSAVANCE 5600 (N=254) | Referred-Care (N=258)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 13 (14)
Urinary Tract Infection (Infections and infestations) | 12 (12) | 14 (18)
Contusion (Injury, poisoning and procedural complications) | 13 (21) | 14 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (24) | 21 (23)
Back Pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 21 (22)
Dizziness (Nervous system disorders) | 9 (10) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts,or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.